CLINICAL TRIAL: NCT00965783
Title: Predictors of the Metabolic Effect of Sleep Loss
Acronym: SDBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: #15207A; 1 RO1 IIL075025
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Apnea; Obstructive Sleep Apnea (OSA); Obesity
Keywords: Sleep, Apnea, OSA, obese, middle-aged
MeSH Terms: conditions — Apnea; Sleep Apnea, Obstructive; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Sleep time restriction
  Interventions: Other: Restriction
- 2 (Experimental): Sleep time extension
  Interventions: Other: Extension

INTERVENTIONS:
Other: Restriction — Time in bed for each subject is restricted by two hours per night for 4 nights
  Arms: 1
Other: Extension — Bedtime is extended by 2 hours per night for 4 nights
  Arms: 2

SUMMARY:
To test whether baseline levels of slow wave activity (SWA) during sleep are lower in obese adults, and even lower in persons with sleep disordered breathing (SDB) compared to lean adults.

To compare levels of SWA in individuals in relation to their sleep time, blood pressure, heart rate, and markers of glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* healthy,
* normal sleepers,
* lean, overweight,
* obese,
* pre menopausal

Exclusion Criteria:

* no shift workers or night-shift workers,
* no mental health disorders,
* no acute or chronic health conditions (stable, well controlled hypertension are accepted),
* no hormonal treatments,
* no substances that may interfere with sleep,
* problems with sleep

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Correlation between SWA, sleep duration,sleep architecture, and biomarkers of the metabolic syndrome in lean, obese with and without obstructive sleep apnea. | study completion

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Chicago, Chicago, Illinois, United States